CLINICAL TRIAL: NCT06088641
Title: Prognostic Impact of Preoperative B-type Natriuretic Peptide for Predicting Myocardial Injury After Non-cardiac Surgery in Patients Who Underwent Open Repair for Abdominal Aortic Aneurysm: a Retrospective Study
Brief Title: Preoperative BNP and MINS in AAA Open Repair
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Yeon Ham, professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0187
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Myocardial Injury After Non-cardiac Surgery
Keywords: AAA; MINS; BNP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower BNP: preoperative Lower BNP
  Interventions: Diagnostic Test: preoperative BNP value
- Higher BNP: preoperative higher BNP
  Interventions: Diagnostic Test: preoperative BNP value

INTERVENTIONS:
Diagnostic Test: preoperative BNP value — preoperative BNP value

SUMMARY:
The aim of this study was to investigate whether preoperative B-type natriuretic peptides serves as an independent predictor of myocardial injury after non-cardiac surgery (MINS) in abdominal aortic aneurysm open repair.

DETAILED DESCRIPTION:
The incidence of MINS was compared between the lower BNP and higher BNP groups, and a stepwise logistic regression analysis was performed to evaluate the predictors for MINS.

ELIGIBILITY:
Inclusion Criteria:

patients who underwent open repair with AAA from September 2010 to October 2021

Exclusion Criteria:

1. Ruptured AAA
2. Traumatic aortic injury
3. Absence of troponin-T value within 30 days of surgery
4. Diagnosis of elevation of troponin-T due to non-ischemic cause (ex: sepsis, pulmonary embolism, atrial fibrillation, cardioversion, etc.)
5. Insufficient medical records

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent AAA open repair
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-07-06 (Estimated)

PRIMARY OUTCOMES:
MINS | 30 days after surgery
  MINS is defined as an elevated Troponin-T within 30 days of surgery. The patients were divided into two groups based on their preoperative BNP levels, and the incidence of MINS was compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam severance Hospital, Seoul, South Korea